CLINICAL TRIAL: NCT05633108
Title: A Retrospective Observational Study Based on the French National Health Insurance Database to Describe Antipsychotic Monotherapy and Polypharmacy Use, Including Loxapac, and to Investigate Their Association With Psychiatric Rehospitalization in Patients With Psychotic Disorders
Brief Title: A Study Based on the French National Health Insurance Database in Participants With Psychotic Disorders
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: LOX-M033-501
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Psychotic Disorders
Keywords: Schizophrenia; Schizotypal disorders; Schizoaffective disorders; Persistent or acute or induced or non-organic delusional disorders; Recurrent depressive disorder
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Depressive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants diagnosed with psychotic disorder at any time between 1 January 2014 and 31 December 2020 and have data available in French nationwide healthcare data system (SNDS) database during this period will be observed retrospectively.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention will be administered.

SUMMARY:
The primary purpose of the study is to compare therapy with antipsychotic medication (antipsychotic monotherapy or antipsychotic combination) versus no antipsychotic medication, and antipsychotic monotherapy versus antipsychotic combination, regarding time to psychiatric rehospitalization, in participants with a psychotic disorder (that is, schizophrenia, schizotypal disorders, schizoaffective disorders, persistent or acute or induced or non-organic delusional disorders, recurrent depressive disorder with psychotic symptoms).

ELIGIBILITY:
Inclusion Criteria:

* At least one discharge for psychiatric hospitalization with a diagnosis of a psychotic disorder between January 1, 2014 and December 31, 2020.
* At least one long-term disease record (LTD), (which is a French administrative status allowing the full reimbursement of the cost of a chronic pathology) with a diagnosis of a psychotic disorder between January 1, 2014 and December 31, 2020.
* Age of 18 years or older at index date (first date found in the previous conditions).

Exclusion Criteria:

• Due to data management constraint, the participants with multiple or temporary identifiers in the database (indistinguishable in database) will be excluded. This happens with twins or migrants, for example.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants hospitalized with a diagnosis of a psychotic disorder will be included in this study at any time between 1 January 2014 and 31 December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 579728 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Time from Discharge from a Psychiatric Hospitalization to the Next Psychiatric Rehospitalization | From 1 January 2014 to 31 December 2020
  Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.

SECONDARY OUTCOMES:
Percentage of Participants Using Loxapac as Monotherapy or With Other Antipsychotic Polypharmacy Medication | From 1 January 2014 to 31 December 2020
  Percentage of participants will be reported using Loxapac or other polypharmacy medications, including anti-psychotic medication (typical/atypical); anti-depressants; anti-psychotic medication sedatives (other than benzodiazepines and z-drugs) and with benzodiazepines and z-drugs; anti-psychotic medication and lithium; anti-psychotic medication mood stabilizers; and with at least one other concomitant medication and without concomitant medication. Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Number of Participants With Consultations Based on a Hospital Psychiatrists, General Practitioner, Private Psychiatric Practitioner or Other Private Specialist | From 1 January 2014 to 31 December 2020
  Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Number of Participants With Hepatic, Glycaemia, Cardiovascular, Lipidic Anomalies Assessments | From 1 January 2014 to 31 December 2020
  Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Number of Participants With Loxapac Treatment Episodes | From 1 January 2014 to 31 December 2020
  Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Number of Participants With Off-drug Loxapac Treatment Period | From 1 January 2014 to 31 December 2020
  The off-drug period is defined as the period between two sequences of Loxapac treatment. Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Duration of Loxapac Treatment | From 1 January 2014 to 31 December 2020
  The time between the start of each Loxapac sequence since the end of Loxapac sequence, switch to another treatment or end of follow-up. Several sequences may exist for one participant. This outcome will be based on medical possession ratio (MPR). MPR will be calculated using B/D formula. Where, B is number of days of supply of Loxapac and D is number of days between the initiation of Loxapac and the end of follow-up. Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Percentage of Days Covered (PDC) With Loxapac Treatment | From 1 January 2014 to 31 December 2020
  PDC will be calculated using A/D formula. Where A is number of days "covered", that is, number of days of supply of Loxapac without carry-over of overlap days and D is number of days between the initiation of Loxapac and the end of follow-up. Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Medical Possession Ratio (MPR) | From 1 January 2014 to 31 December 2020
  MPR will be calculated using B/D formula. Where, B is number of days of supply of Loxapac and D is number of days between the initiation of Loxapac and the end of follow-up. Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Fixed Medical Possession Ratio (FMPR) | From 1 January 2014 to 31 December 2020
  FMPR will be evaluated using MPR and PDC. MPR will be calculated using B/D formula. Where, B is number of days of supply of Loxapac and D is number of days between the initiation of Loxapac and the end of follow-up. PDC will be calculated using A/D formula. Where A is number of days "covered", that is, number of days of supply of Loxapac without carry-over of overlap days and D is number of days between the initiation of Loxapac and the end of follow-up. Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Number of Participants Categorized Based on all Hospitalizations, Psychiatric and Other Hospitalizations | From 1 January 2014 to 31 December 2020
  Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Number of Participants With Passage Through Emergency Department of Hospital | From 1 January 2014 to 31 December 2020
  Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Number of Participants Using Different Antipsychotic Medications | From 1 January 2014 to 31 December 2020
  The different antipsychotic medication (other than Loxapac) among the following categories: clozapine, olanzapine, aripiprazole, risperidone, quetiapine, amisulpride, others oral medication. Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Cumulative Duration of Loxapac as Monotherapy | From 1 January 2014 to 31 December 2020
  Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Cumulative Duration of an Atypical/Typical Antipsychotic Drug Taken as Monotherapy Other Than Loxapac | From 1 January 2014 to 31 December 2020
  Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Cumulative Duration of Anti-Psychotic Biotherapy | From 1 January 2014 to 31 December 2020
  Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Cumulative Duration of Loxapac and an Atypical/Typical Antipsychotic Therapy | From 1 January 2014 to 31 December 2020
  Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Cumulative Duration of Other Antipsychotic Polypharmacy | From 1 January 2014 to 31 December 2020
  Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.
Cumulative Duration of Periods Without any Antipsychotic Treatment | From 1 January 2014 to 31 December 2020
  Participants will be censored in case of death or lost to follow up or on 31 Dec 2020, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Eisai Ltd. European Knowledge Centre, Hatfield, Hertfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.